CLINICAL TRIAL: NCT06109974
Title: Evaluation of an Algorithm That Can Detect COPD by Intelligent Terminal Device
Brief Title: Evaluate the Accuracy of a COPD Screening Algorithm Model
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Collaborators: Civil Aviation General Hospital (Other); Shichahai Community Health Service Center of Xicheng District Beijing (Unknown); The Hospital of Changping District Beijing (Unknown); Baizhifang Community Health Service Center of Xicheng District Beijing (Unknown)
Responsible Party: Principal Investigator, Guangfa Wang, Prof. & MD., Peking University First Hospital
Other Study IDs: 2022083-20230810
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: COPD
Keywords: COPD; Intelligent Terminal Device; Algorithm model
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with high risk of COPD: no intervention

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is one of the most common respiratory diseases. Early detection and treatment are critical to prevent the deterioration of COPD. In this study, we have established an algorithm that can detect and infer the severity of COPD from physiological parameters and audio data collected by wearable devices, and in this stage, we aim to evaluate the accuracy of this algorithm.

DETAILED DESCRIPTION:
The investigators have established an algorithm that can detect COPD from physiological parameters, coughing sounds, and forceful expiratory sounds collected by wearable devices. This study will test the accuracy of this algorithm.

In this study, 404 residents at high risk of COPD (COPD-PS score≥5) will be enrolled. Questionnaires related to COPD will be collected, subjects will undergo pulmonary function tests and electrocardiogram. Physiological parameters such as oxygen saturation and heart rate will be collected by a wearable device 3 times for 2 minutes each time, and coughing sound will be collected. As spirometry is the gold standard for the diagnosis of COPD, the accuracy of COPD diagnosis algorithm model by intelligent terminal devices will be verified.

The study protocol has been approved by the Peking University First Hospital Institutional Review Board (IRB) (2022-083). Any protocol modifications will be submitted for the IRB review and approval.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 18, no gender restrictions.
2. Participants at high risk of COPD (COPD-PS score ≥5).
3. Able to carry out daily activities and wear wearable devices.
4. Willing to participate in the study, willing to comply with the study protocol, and have the ability to sign informed consent.
5. Possess mobile communication equipment, which can meet the requirement of installing wearable device applications and recording function.

Exclusion Criteria:

1. Diagnosed with chronic respiratory diseases other than COPD, such as asthma, lung cancer, active tuberculosis, bronchiectasis and diffuse lung diseases (interstitial pneumonia, occupational lung disease, sarcoidosis, etc.).
2. lobectomy and/or lung transplantation, pleural disease.
3. Complicated with serious underlying diseases, including severe mental illness, intellectually impaired diseases, neurological disease (resulting in limb movement disorder), malignant tumor (PS score > 2), chronic liver disease (transaminase > 3 times the upper limit of normal), heart failure (NYHA> Grade 3), autoimmune disease, chronic kidney disease (CKD-5), unstable coronary artery disease, arrhythmia (atrial fibrillation, atrial flutter, severe ventricular arrhythmia), congenital heart disease, pulmonary hypertension, etc., or life expectancy of less than 6 months.
4. Malnutrition (BMI<18 kg/m2).
5. Bilateral wrist and hand edema, wrist soft tissue injury, inability to wear a watch/bracelet due to incomplete skin.
6. Dual upper limb pigmentation or abnormal blood supply (occlusion, thrombosis, trauma, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participants at high risk of COPD
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
The diagnostic accuracy of the algorithm for COPD | 1 year
  The diagnostic accuracy of the algorithm for COPD

SECONDARY OUTCOMES:
The diagnostic sensitivity and specificity of the algorithm | 1 year
  The diagnostic sensitivity and specificity of the algorithm
The diagnostic accuracy of COPD-PS score for COPD | 1 year
  The diagnostic accuracy of COPD-PS score for COPD

CONTACTS AND LOCATIONS:
Overall Officials: Guangfa Wang, MD, Study Chair — Peking University First Hospital
Locations (5):
- China (5):
  - Baizhifang Community Health Service Center of Xicheng District Beijing, Beijing, Beijing Municipality
  - Civil Aviation General Hospita, Beijing, Beijing Municipality
  - Guangfa Wang, Beijing, Beijing Municipality
  - Shichahai community health service center, Beijing, Beijing Municipality
  - The Hospital of Changping District Beijing, Beijing, Beijing Municipality